CLINICAL TRIAL: NCT02432846
Title: An Open-label, Randomized, Controlled, Multicenter, Phase II Study Evaluating Safety and Efficacy of Intratumorally Administered Intuvax Pre-nephrectomy Followed by Sunitinib Post-nephrectomy, Compared to Sunitinib Post-nephrectomy in Metastatic Renal Cell Carcinoma Patients
Brief Title: Intratumoral Vaccination With Intuvax Pre-nephrectomy Followed by Sunitinib Post-nephrectomy vs Sunitinib Post-nephrectomy in Newly Diagnosed Metastatic Renal Cell Carcinoma (mRCC)
Acronym: MERECA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mendus (Industry)
Collaborators: TFS Trial Form Support (Industry); Accelovance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM-201; 2014-004510-28 (EudraCT Number)
Record Dates: First submitted 2015-04-15; First posted 2015-05-04 (Estimated); Results first posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-07

CONDITIONS: Renal Cell Carcinoma, Metastatic
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intuvax (INN: ilixadencel)+ Nephrectomy+Sunitinib (Experimental): Two Intuvax (INN: ilixadencel) doses (10 million cells/dose) 14 days apart before nephrectomy, followed by Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Interventions: Biological: Intuvax (INN: ilixadencel); Drug: Sunitinib
- Nephrectomy+Sunitinib (Active Comparator): Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Biological: Intuvax (INN: ilixadencel) — Therapeutic dose (10 million cells/dose): allogeneic, pro-inflammatory dendritic cells.
  Other Names: COMBIG-DC
  Arms: Intuvax (INN: ilixadencel)+ Nephrectomy+Sunitinib
Drug: Sunitinib — Cytostatic/cytotoxic drug: protein kinase inhibitor .
  Other Names: Sutent

SUMMARY:
The purpose of this study is to compare tumor response, progression free survival (PFS) and overall survival (OS) in newly diagnosed mRCC patients treated with Intuvax (INN: ilixadencel) pre-nephrectomy followed by Sunitinib post-nephrectomy vs Sunitinib post-nephrectomy patients.

DETAILED DESCRIPTION:
Patients, all planned for nephrectomy, will be stratified according to the Heng risk criteria (high risk patients vs. intermediate risk patients) and randomized in a 2:1 ratio to receive Intuvax (INN: ilixadencel)+ Sunitinib or Sunitinib alone.

Two doses of Intuvax (INN: ilixadencel) will be administered in to the primary tumour before nephrectomy. The control group will be scheduled for nephrectomy directly.

All patients will start Sunitinib treatment 5-8 weeks after operation.

Results from the phase I study, together with the results reported in the literature on the use of autologous dendritic cells (DCs) in combination with Sunitinib encourage Immunicum aktiebolag (AB) to further investigate the possibility of exploiting Intuvax (INN: ilixadencel) 10 million cells/dose when combined with Sunitinib for the treatment of mRCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Newly (<6 months) diagnosed RCC (histological/cytological verification is optional) with at least one (1) CT-verified metastasis ≥10mm for which complete metastasectomy is not planned. US patients must have verified clear-cell tumor histology
2. Planned resection of primary tumor
3. Primary tumor diameter ≥40 mm
4. Candidate for first-line therapy with sunitinib initiated 5-8 weeks after nephrectomy
5. Female or male ≥18 years of age
6. Willing and able to provide informed consent
7. Adequate hematological parameters, i.e:

   * B-Leukocyte count ≥4.5 x10e9/L
   * B-Platelet count ≥150 x10e9/L
   * B-Hemoglobin ≥90 g/L
8. S-creatinine and S-bilirubin ≤ 1.5 x upper limit of normal (ULN). Serum alanine aminotransferase (S-ALAT) and serum aspartate aminotransferase (S-ASAT) ≤ 2.5 x ULN (or ≤5 in case of liver metastases)
9. Female who has been post-menopausal for more than one (1) year or female of childbearing potential agreeing to use a highly efficient method of contraception (i.e. a method with less than 1% failure rate [e.g. sterilization, hormone implants, hormone injections, some intrauterine devices, or vasectomized partner or combined birth control pills]) Female of childbearing potential must have a negative from Screening until 90 days after last dose of Intuvax and/or until completed sunitinib treatment whichever occurs later.blood pregnancy test at Screening, and if randomized to vaccination a negative blood or urine pregnancy test within one (1) day before each dose of Intuvax) and must not be lactating.

or Male agreeing to use condoms from Screening until 90 days after last dose of Intuvax and/or until completed sunitinib treatment whichever occurs later, or male having a female partner who is using a highly efficient method of contraception as described above.

Exclusion Criteria:

1. Life expectancy less than 4 months
2. Central nervous system (CNS) metastasis that is symptomatic or progressing or untreated or that required current therapy (e.g. evidence of new or enlarging CNS metastasis or new neurological symptoms attributable to CNS metastases)
3. Active autoimmune disease which requires treatment with systemic immunosuppressive agents, e.g. inflammatory bowel disease, multiple sclerosis, sarcoidosis, psoriasis, autoimmune hemolytic anemia, rheumatoid arthritis, systemic lupus erythematosus (SLE), vasculitis, Sjögren's syndrome, scleroderma, autoimmune hepatitis, and other rheumatological diseases
4. Treatment with per oral systemic corticosteroids exceeding 10mg/day within seven (7) days before Screening until nephrectomy (inhaled, intranasal and local steroids accepted irrespective of dose)
5. Known cardiomyopathy and/or clinical significant abnormal ECG findings at Screening disqualifying the patient from nephrectomy and from subsequent sunitinib treatment
6. Karnofsky performance status <70%
7. National Cancer Institute (NCI) Common Terminology criteria for Adverse Events (CTCAE) Grade 3 hemorrhage within 28 days before Screening
8. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication
9. Clinically significant gastrointestinal abnormalities
10. Uncontrolled hypertension, or uncontrolled diabetes mellitus
11. Pulmonary embolism within 12 months before screening
12. Prior history of invasive cancer within 5 years before screening, except for adequately treated in situ carcinomas or non-melanoma skin cancer
13. Ongoing infection that requires parenteral treatment with antibiotics
14. Active or latent virus disease (HIV, hepatitis B and hepatitis C)
15. Eastern Cooperative Oncology Group (ECOG) performance status >2 after optimization of analgesics
16. Abnormal and clinical significant coagulation parameters at the discretion of the Investigator, i.e.:

    * Prothrombin Time - International Normalized Ratio (PT-INR)
    * Activated Partial Thromboplastin Time (APTT) patients being treated with anticoagulants are excluded if the coagulation parameters are outside the therapeutic intervals as described in the summary of product characteristics (SmPC) / United States prescribing information (USPI) for the administered treatment
17. Known major adverse reaction/event in connection with previously made vaccination (e.g. asthma, anaphylaxis or other serious reaction)
18. Known hypersensitivity or allergy sunitinib or to chemically related products or likely to be exacerbated to by any component of the study products
19. Prior systemic antitumour therapy within 28 days before Screening Visit. However, local radiation therapy to any area except for the abdominal/retroperitoneal area including the kidney tumour is allowed
20. Exposure to other investigational products within 28 days prior to Screening Visit
21. patients on anticoagulants for whom temporarily stop and start, supported by low molecular weight heparin (or other anticoagulation therapy at the discretion of the investigator and or per local standard of care) during vaccination and nephrectomy, is not an option
22. History of alcohol or substance abuse
23. Any reason that, in the opinion of the Investigator, contraindicates that the patient participates in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-04; Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Börje Ljungberg, MD, Prof, Principal Investigator — Umeå University Hospital
Locations (28):
- United States (5):
  - University of Illinois, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Health Partners Institute, Saint Paul, Minnesota
  - Duke Cancer Institute, Durham, North Carolina
- University Hospital Olomouc, Olomouc, Czechia
- France (2):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Universitaire de Toulouse-Hôpital Rangueil, Toulouse
- Hungary (2):
  - University of Debrecen, Debrecen
  - Szent-Györgyi Albert Klinikai Központ, Szeged
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
- Poland (4):
  - Niepubliczny Zakład Opieki Zdrowotnej Vesalius Sp. z o.o., Krakow
  - Wojewodzki Szpital Specjalistyczny, Lublin
  - Military Institute of Medicine, Warsaw
  - Mazowiecki Szpital Onkologiczny, Wieliszew
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitari Parc Tauli, Sabadell
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Huddinge
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
- United Kingdom (2):
  - The Churchill Hospital, Oxford
  - Royal Preston Hospital, Preston

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient's first visit was 28 April 2015 and last patient's last visit was 17 June 2019. Patients were recruited from Sweden (n=31), France (n=4), United States (n=2), Czech Republic (n=6), Latvia (n=6), Poland (n=12), Spain (n=18), Hungary (n=5), United Kingdom (n=4).
Pre-assignment Details: 117 patients with newly diagnosed metastatic renal cell cancer were screened according to the inclusion and exclusion criteria. The 88 eligible patients were randomized to either of two treatments: Intuvax (INN: ilixadencel) + Sunitinib or Sunitinib-only. Patients were stratified according to Heng criteria, as either high-risk or intermediate-risk. Results are presented by risk stratum and treatment (4 groups) and by treatment overall (2 groups), i.e. the 6 groups are not mutually exclusive.
Groups:
- Intuvax (INN: Ilixadencel)+ Nephrectomy+ Sunitinib: High-risk Stratum: Two Intuvax (INN: ilixadencel) doses (10 million cells/dose) 14 days apart before nephrectomy, followed by Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Intuvax (INN: ilixadencel): Therapeutic dose (10 million cells/dose): allogeneic, pro-inflammatory dendritic cells.
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  High-risk stratum.
- Nephrectomy + Sunitinib: High-risk Stratum: Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  High-risk stratum.
- Intuvax (INN Ilixadencel)+ Nephrectomy+Sunitinib: Intermediate-risk Stratum: Two Intuvax (INN: ilixadencel) doses (10 million cells/dose) 14 days apart before nephrectomy, followed by Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Intuvax (INN: ilixadencel): Therapeutic dose (10 million cells/dose): allogeneic, pro-inflammatory dendritic cells.
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  Intermediate-risk stratum.
- Nephrectomy + Sunitinib: Intermediate-risk Stratum: Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  Intermediate-risk stratum.
- Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: Total: Two Intuvax (INN: ilixadencel) doses (10 million cells/dose) 14 days apart before nephrectomy, followed by Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Intuvax (INN: ilixadencel): Therapeutic dose (10 million cells/dose): allogeneic, pro-inflammatory dendritic cells.
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  High risk and intermediate risk strata combined.
- Nephrectomy+Sunitinib: Total: Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  High-risk and intermediate-risk strata combined.
Period: Overall Study (4 Arms/Strata)
Arm/Group | Intuvax (INN: Ilixadencel)+ Nephrectomy+ Sunitinib: High-risk Stratum | Nephrectomy + Sunitinib: High-risk Stratum | Intuvax (INN Ilixadencel)+ Nephrectomy+Sunitinib: Intermediate-risk Stratum | Nephrectomy + Sunitinib: Intermediate-risk Stratum | Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: Total | Nephrectomy+Sunitinib: Total
Started | 17 | 8 | 41 | 22 | 0 | 0
Completed | 2 | 0 | 17 | 8 | 0 | 0
Not Completed | 15 | 8 | 24 | 14 | 0 | 0
Not completed — Death | 3 | 2 | 4 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Other (reason not specified) | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Disease progression | 8 | 5 | 15 | 9 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Period: Overall Study (2 Total/Combined Groups)
Arm/Group | Intuvax (INN: Ilixadencel)+ Nephrectomy+ Sunitinib: High-risk Stratum | Nephrectomy + Sunitinib: High-risk Stratum | Intuvax (INN Ilixadencel)+ Nephrectomy+Sunitinib: Intermediate-risk Stratum | Nephrectomy + Sunitinib: Intermediate-risk Stratum | Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: Total | Nephrectomy+Sunitinib: Total
Started | 0 | 0 | 0 | 0 | 58 | 30
Completed | 0 | 0 | 0 | 0 | 19 | 8
Not Completed | 0 | 0 | 0 | 0 | 39 | 22
Not completed — Death | 0 | 0 | 0 | 0 | 7 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Other (reason not specified) | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Disease progression | 0 | 0 | 0 | 0 | 23 | 14
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The 6 groups are not mutually exclusive. The patients are presented both separately by risk stratum and treatment (4 groups) and by treatment group overall (2 groups) where high-risk and intermediate-risk strata are combined. This split of baseline characteristics provides transparency for efficacy outcomes that are analysed by these 6 groups.
Groups:
- Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: High-risk Stratum: Two Intuvax (INN: ilixadencel) doses (10 million cells/dose) 14 days apart before nephrectomy, followed by Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Intuvax (INN: ilixadencel): Therapeutic dose (10 million cells/dose): allogeneic, pro-inflammatory dendritic cells.
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  High-risk stratum.
- Nephrectomy+Sunitinib: High-risk Stratum: Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  High-risk stratum.
- Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: Intermediate-risk Stratum.: Two Intuvax (INN: ilixadencel) doses (10 million cells/dose) 14 days apart before nephrectomy, followed by Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Intuvax (INN: ilixadencel): Therapeutic dose (10 million cells/dose): allogeneic, pro-inflammatory dendritic cells.
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  Intermediate-risk stratum.
- Nephrectomy+Sunitinib: Intermediate-risk Stratum: Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  Intermediate-risk stratum.
- Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: Total: Two Intuvax (INN: ilixadencel) doses (10 million cells/dose) 14 days apart before nephrectomy, followed by Sunitinib treatment post-nephrectomy according to clinical practice until RECIST verified progressive disease or End-of-Study (78 weeks after screening).
  Intuvax (INN: ilixadencel): Therapeutic dose (10 million cells/dose): allogeneic, pro-inflammatory dendritic cells.
  Sunitinib: Cytostatic/cytotoxic drug: protein kinase inhibitor.
  High-risk and intermediate-risk strata combined.
- Total: Total of all reporting groups
Arm/Group | Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: High-risk Stratum | Nephrectomy+Sunitinib: High-risk Stratum | Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: Intermediate-risk Stratum. | Nephrectomy+Sunitinib: Intermediate-risk Stratum | Intuvax (INN: Ilixadencel)+ Nephrectomy+Sunitinib: Total | Nephrectomy+Sunitinib: Total | Total
Number analyzed (Participants) | 17 | 8 | 41 | 22 | 58 | 30 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Screening Visit Population: The patients are presented both separately by risk stratum and treatment (4 groups) and by treatment group overall (2 groups) where high-risk and intermediate-risk strata are combined. This split of baseline characteristics provides transparency for efficacy outcomes that are analysed by these 6 groups.
  years
    Age (4 arms/strata): number analyzed (Participants) | 17 | 8 | 41 | 22 | 0 | 0 | 88
    Age (4 arms/strata) | 62.0 (9.6) | 60.5 (7.7) | 61.0 (8.4) | 65.5 (10.3) |  |  | 62.3 (9.1)
    Age (2 total/combined groups): number analyzed (Participants) | 0 | 0 | 0 | 0 | 58 | 30 | 88
    Age (2 total/combined groups) |  |  |  |  | 61.3 (8.7) | 64.2 (9.8) | 62.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The patients are presented both separately by risk stratum and treatment (4 groups) and by treatment group overall (2 groups) where high-risk and intermediate-risk strata are combined. This split of baseline characteristics provides transparency for efficacy outcomes that are analysed by these 6 groups.
  Participants
    Sex (4 arms/strata): number analyzed (Participants) | 17 | 8 | 41 | 22 | 0 | 0 | 88
    Sex (4 arms/strata): Female | 2 | 2 | 11 | 7 | 0 | 0 | 22
    Sex (4 arms/strata): Male | 15 | 6 | 30 | 15 | 0 | 0 | 66
    Sex (2 total/combined groups): number analyzed (Participants) | 0 | 0 | 0 | 0 | 58 | 30 | 88
    Sex (2 total/combined groups): Female | 0 | 0 | 0 | 0 | 13 | 9 | 22
    Sex (2 total/combined groups): Male | 0 | 0 | 0 | 0 | 45 | 21 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The patients are presented both separately by risk stratum and treatment (4 groups) and by treatment group overall (2 groups) where high-risk and intermediate-risk strata are combined. This split of baseline characteristics provides transparency for efficacy outcomes that are analysed by these 6 groups.
  Participants
    race (4 arms/strata): number analyzed (Participants) | 17 | 8 | 41 | 22 | 0 | 0 | 88
    race (4 arms/strata): American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    race (4 arms/strata): Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    race (4 arms/strata): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    race (4 arms/strata): Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    race (4 arms/strata): White | 16 | 6 | 41 | 22 | 0 | 0 | 85
    race (4 arms/strata): More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    race (4 arms/strata): Unknown or Not Reported | 1 | 2 | 0 | 0 | 0 | 0 | 3
    Race (2 total/combined groups): number analyzed (Participants) | 0 | 0 | 0 | 0 | 58 | 30 | 88
    Race (2 total/combined groups): American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race (2 total/combined groups): Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race (2 total/combined groups): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race (2 total/combined groups): Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race (2 total/combined groups): White | 0 | 0 | 0 | 0 | 57 | 28 | 85
    Race (2 total/combined groups): More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Race (2 total/combined groups): Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) - Days (FAS)
Description: OS is the time from randomization until date of death. The patients who were alive at the end of study were followed for survival status (alive/date of death) through medical records, databases and public records according to the time frame below.
  Due to censored data, estimates of upper 95% CI could not be determined in all reporting groups.
Time Frame: From the randomization to the date of death, up to 5 years after the last participant's 18-month survival data.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Intuvax (INN: Ilixadencel) + Sunitinib, High-risk: Intuvax (INN: ilixadencel) + sunitinib, high-risk stratum
- Sunitinib-only, High-risk: Sunitinib-only, high-risk stratum
- Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk: Intuvax (INN: ilixadencel) + sunitinib, intermediate-risk stratum
- Sunitinib-only, Intermediate-risk: Sunitinib-only, intermediate-risk stratum
- Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata): Intuvax (INN: ilixadencel) + sunitinib, high and intermediate risk strata combined
- Sunitinib-only, Total (Both Strata): Sunitinib-only, high and intermediate risk strata combined
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 16 | 8 | 40 | 22 | 56 | 30
days | 323 [152 to 682] | 282 [39 to NA] — Upper 95% CI not reached due to censored data. | 1270 [852 to NA] — Upper 95% CI not reached due to censored data. | 1099 [234 to 1368] | 1082 [432 to NA] — Upper 95% CI not reached due to censored data. | 770 [234 to 1241]
Statistical Analysis 1: Comparison: Intuvax (INN: Ilixadencel) + Sunitinib, High-risk vs Sunitinib-only, High-risk; Test type: Other — Exploratory superiority (non-powered); p = 0.964, Log Rank; Hazard Ratio (HR) = 0.978, 95% CI 2-sided [0.371 to 2.579]
Statistical Analysis 2: Comparison: Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk vs Sunitinib-only, Intermediate-risk; Test type: Other — Exploratory superiority (non-powered); p = 0.163, Log Rank; Hazard Ratio (HR) = 0.619, 95% CI 2-sided [0.314 to 1.222]
Statistical Analysis 3: Comparison: Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) vs Sunitinib-only, Total (Both Strata); Test type: Other — Exploratory superiority (non-powered); p = 0.250, Log Rank; Hazard Ratio (HR) = 0.732, 95% CI 2-sided [0.421 to 1.270]

2. Primary Outcome: Overall Survival - Days (PPS)
Description: OS is the time from randomization until date of death. The patients who were alive at the end of study were followed for survival status (alive/date of death) through medical records, databases and public records according to the time frame below.
  Due to censored data, upper 95% CI could not be determined in all reporting groups.
Time Frame: From the randomization to the date of death, up to 5 years after the last patient's 18-month survival data.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata): Intuvax (INN: ilixadencel) + sunitinib, high and intermediate-risk strata combined
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 12 | 8 | 34 | 19 | 46 | 27
days | 352 [240 to NA] — Upper 95% CI not reached due to censored data. | 282 [39 to NA] — Upper 95% CI not reached due to censored data. | 1745 [911 to NA] — Upper 95% CI not reached due to censored data. | 1185 [678 to NA] — Upper 95% CI not reached due to censored data. | 1265 [684 to NA] — Upper 95% CI not reached due to censored data. | 1024 [342 to 1368]
Statistical Analysis 1: Comparison: Intuvax (INN: Ilixadencel) + Sunitinib, High-risk vs Sunitinib-only, High-risk; Test type: Other — Exploratory superiority (non-powered); p = 0.596, Log Rank; Hazard Ratio (HR) = 0.756, 95% CI 2-sided [0.268 to 2.134]
Statistical Analysis 2: Comparison: Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk vs Sunitinib-only, Intermediate-risk; Test type: Other — Exploratory superiority (non-powered); p = 0.285, Log Rank; Hazard Ratio (HR) = 0.661, 95% CI 2-sided [0.308 to 1.418]
Statistical Analysis 3: Comparison: Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) vs Sunitinib-only, Total (Both Strata); Test type: Other — Exploratory superiority (non-powered); p = 0.240, Log Rank; Hazard Ratio (HR) = 0.699, 95% CI 2-sided [0.378 to 1.290]

3. Primary Outcome: 18-Months' Overall Survival Percentage (FAS)
Description: The 18-month survival percentage was defined as the percentage of patients alive 18 months after randomization.
Time Frame: At 18 months (544 days)
Measure: Number; unit: Percentage of participants
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 16 | 8 | 40 | 22 | 56 | 30
Percentage of participants | 30 | 38 | 77 | 76 | 63 | 66
Statistical Analysis 1: Comparison: Intuvax (INN: Ilixadencel) + Sunitinib, High-risk vs Sunitinib-only, High-risk vs Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk vs Sunitinib-only, Intermediate-risk; Test type: Other — Exploratory superiority (non-powered); p = 0.812, Log Rank

4. Primary Outcome: 18-Months' Overall Survival Percentage (PPS)
Description: The 18-month survival percentage was defined as the percentage of patients alive 18 months after randomization.
Time Frame: At 18 months (544 days)
Measure: Number; unit: Percentage of participants
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 12 | 8 | 34 | 19 | 46 | 27
Percentage of participants | 31 | 38 | 82 | 84 | 68 | 70
Statistical Analysis 1: Comparison: Intuvax (INN: Ilixadencel) + Sunitinib, High-risk vs Sunitinib-only, High-risk vs Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk vs Sunitinib-only, Intermediate-risk; Test type: Other — Exploratory superiority (non-powered); p = 0.861, Log Rank

5. Secondary Outcome: Progression Free Survival (PFS) From Start of Sunitinib According to RECIST 1.1.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by radiographic assessment: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  Due to the large amount of censored data, estimates of median and/or a 95% CI could not be reliably determined in all reporting groups.
  Baseline data are reported for the safety data set (all patients randomized) whereas PFS is analyzed for the full analysis set (FAS). Two patients in the safety data set were not included in the FAS since they withdrew prior to start of treatment.
Time Frame: From Sunitinib-Start to progressive disease or death, up to 18 months.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Sunitinib-only High-risk: Sunitinib-only, high-risk stratum
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 13 | 6 | 33 | 19 | 46 | 25
days | 254 [43 to NA] — Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined. | NA [NA to NA] — Due to the large amount of censored data, estimates of median and 95% CI could not be reliably determined. | 478 [249 to NA] — Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined. | 417 [149 to NA] — Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined. | 360 [249 to NA] — Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined. | 337 [149 to NA] — Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined.

6. Secondary Outcome: Objective Response Rate (ORR) From Start of Sunitinib Treatment and Duration of Response in Each Subgroup.
Description: Objective response rate was defined as the percentage of patients with complete response (CR) and partial response (PR).Tumor response was evaluated centrally according to the RECIST 1.1 guideline.
Time Frame: From start of sunitinib treatment up to 18 months
Measure: Number; unit: Percentage of participants
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 13 | 6 | 32 | 19 | 45 | 25
Percentage of participants | 38.5 | 66.7 | 46.9 | 42.1 | 44.4 | 48.0

7. Secondary Outcome: Number of Participants With Specific Best Overall Response
Description: The best overall response is the best response recorded from the start of the treatment sunitinib until disease progression/recurrence; taking as reference for progressive disease (PD) the smallest measurements recorded since the treatment started. In general, the patient's best response assignment depended on the achievement of the measurement criteria.
Time Frame: From start of sunitinib treatment up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 13 | 6 | 32 | 19 | 45 | 25
Participants
  Complete Response (CR) | 1 | 0 | 4 | 1 | 5 | 1
  Partial Response (PR) | 4 | 4 | 11 | 7 | 15 | 11
  Progressive Disease (PD) | 4 | 0 | 3 | 2 | 7 | 2
  Stable Disease (SD) | 2 | 2 | 13 | 7 | 15 | 9
  Non-CR/Non-PD | 2 | 0 | 0 | 1 | 2 | 1
  No Disease (ND) | 0 | 0 | 1 | 1 | 1 | 1

8. Secondary Outcome: Disease Control Rate
Description: Best overall response (CR, PR or SD) evaluated from Sunitinib-Start for patients with available data.
Time Frame: From start of sunitinib treatment up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 13 | 6 | 32 | 19 | 45 | 25
Participants | 7 | 6 | 28 | 15 | 35 | 21

9. Secondary Outcome: Duration of Response
Description: The duration of response was calculated for only those patients who responded. It was the time from first objective response to first observed progression of disease or death if the death was due to disease progression (whichever came first).
Time Frame: From first date of CR or PR until date of PD or death, up to 18 months.
Measure: Median (Full Range); unit: days
Groups:
- Full Analysis Set (FAS): All patients randomized being evaluable for any high or intermediate stratum related efficacy endpoint.
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata) | Full Analysis Set (FAS)
Number analyzed (Participants) | 5 | 4 | 15 | 8 | 20 | 12 | 32
days | 175.0 [101 to 219] | 81.5 [42 to 126] | 316.0 [1 to 512] | 108.0 [1 to 409] | 215.0 [1 to 512] | 87.0 [1 to 409] | 169.5 [1 to 512]

10. Secondary Outcome: Duration of Clinical Benefit
Description: Disease control rate (DCR) also called Clinical Benefit Rate, was defined as the proportion of patients with CR or PR or SD.
Time Frame: From first date of clinical benefit (CR, PR or SD) until date of PD or death, up to 18 months.
Measure: Median (Full Range); unit: days
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata) | Full Analysis Set (FAS)
Number analyzed (Participants) | 7 | 6 | 28 | 15 | 35 | 21 | 56
days | 212.0 [1 to 434] | 60.0 [1 to 206] | 323.5 [29 to 512] | 295.0 [1 to 451] | 219.0 [1 to 512] | 133.0 [1 to 451] | 211.0 [1 to 512]

11. Secondary Outcome: Duration of Stable Disease
Description: The duration of SD was calculated for only those patients who exhibited a best response of SD response as per RECIST v1.1. It was the time from first SD response to first observed progression of disease or death if the death was due to disease progression (whichever came first), up to 18 months.
Time Frame: From first date of SD until PD or date of death, up to 18 months.
Measure: Median (Full Range); unit: days
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata) | Full Analysis Set (FAS)
Number analyzed (Participants) | 2 | 2 | 13 | 7 | 15 | 9 | 24
days | 63.5 [1 to 126] | 10.5 [1 to 20] | 169.0 [29 to 427] | 210.0 [50 to 449] | 126.0 [1 to 427] | 133.0 [1 to 449] | 129.5 [1 to 449]

12. Secondary Outcome: Time to Progression (TTP)
Description: Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined in all reporting groups.
Time Frame: Time from Sunitinib-Start to date of either PD according to RECIST 1.1 or clinical progression as evaluated by the Investigator, up to 18 months.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 13 | 6 | 33 | 19 | 46 | 25
days | 169 [43 to NA] — Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined. | 143 [48 to 248] | 388 [213 to NA] — Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined. | 417 [93 to NA] — Due to the large amount of censored data, estimate of upper 95% CI could not be reliably determined. | 254 [169 to 478] | 251 [93 to 434]

13. Secondary Outcome: Percentage of Tumor Area With Infiltrating Cluster of Differentiation 8+ (CD8+) T-cells
Description: Relative number of tumor-infiltrating CD8+ T-cells in the resected primary tumor compared to number of infiltrating CD8+ T-cells in available diagnostic pre-biopsy (sample from either primary tumor or metastasis), was not to be evaluated as described in the protocol due to missing pre-biopsy samples). Instead an automated and validated quantification of percentage of CD8+ tissue in delineated tumor area was made.
Time Frame: At resection of primary tumor.
Measure: Median (Full Range); unit: Percentage of tumor area
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata) | Full Analysis Set (FAS)
Number analyzed (Participants) | 14 | 7 | 38 | 20 | 52 | 27 | 79
Percentage of tumor area | 1.0 [0 to 8] | 1.1 [0 to 4] | 1.2 [0 to 13] | 0.8 [0 to 8] | 1.1 [0 to 13] | 0.8 [0 to 8] | 1.1 [0 to 13]

14. Post Hoc Outcome: Confirmed Objective Response Rate
Description: Percentage of patients with the individual's confirmed best overall response scored as CR or PR at least 4 weeks apart from the CT/MRI with the initial best response of CR or PR. Tumor response was evaluated centrally according to the response evaluation criteria in solid tumors (RECIST) 1.1 guideline.
Time Frame: From start of sunitinib treatment up to 18 months
Measure: Number; unit: Percentage of participants
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 13 | 6 | 32 | 19 | 45 | 25
Percentage of participants | 38.5 | 33.3 | 43.8 | 21.1 | 42.2 | 24.0

15. Post Hoc Outcome: Confirmed Best Overall Response
Description: Number of patients with the individual's best overall response at initial CT/MRI confirmed by a best response level at least 4 weeks later in accordance with RECIST 1.1.
Time Frame: From start of sunitinib treatment up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, High-risk | Sunitinib-only, High-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Intermediate-risk | Sunitinib-only, Intermediate-risk | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
Number analyzed (Participants) | 13 | 6 | 32 | 19 | 45 | 25
Participants
  Complete response (CR) | 0 | 0 | 3 | 0 | 3 | 0
  Partial response (PR) | 5 | 2 | 11 | 4 | 16 | 6
  Stable disease (SD) | 1 | 1 | 10 | 9 | 11 | 10
  Missing | 7 | 3 | 8 | 6 | 15 | 9

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from first dose to last follow-up, up to 18 months. All-cause mortality was collected from first dose up to 5 years after last participant's 18-month survival data.
Description: Adverse events are presented overall by treatment, not further split by strata, since the split by strata is deemed to be relevant for efficacy endpoints only.
Arm/Group | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) | Sunitinib-only, Total (Both Strata)
All-Cause Mortality (participants affected / at risk) | 24/58 | 17/30
Serious Adverse Events (participants affected / at risk) | 27/58 | 17/30
Other Adverse Events (participants affected / at risk) | 54/58 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) (N=58) | Sunitinib-only, Total (Both Strata) (N=30)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic bone disease prophylaxis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Recorded as "Metastatic pain"
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 1 (1)
Multi-organ disorder (General disorders) | 0 (0) | 1 (1) — Listed as "Multi-organ failure"
Pyrexia (General disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Post procedural infection (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intuvax (INN: Ilixadencel) + Sunitinib, Total (Both Strata) (N=58) | Sunitinib-only, Total (Both Strata) (N=30)
Asthenia (General disorders) | 11 (19) | 5 (5)
Fatigue (General disorders) | 14 (14) | 8 (11)
General physical health deterioration (General disorders) | 3 (3) | 1 (1)
Mucosal inflammation (General disorders) | 6 (10) | 1 (1)
Pain (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 11 (18) | 4 (6)
Anxiety (Psychiatric disorders) | 5 (6) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Blood creatinine increased (Investigations) | 6 (9) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5) | 4 (4)
Platelet count decreased (Investigations) | 2 (3) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 14 (19) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 3 (4)
Dysgeusia (Nervous system disorders) | 9 (14) | 5 (7)
Headache (Nervous system disorders) | 7 (8) | 1 (1)
Paresis (Nervous system disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 14 (23) | 7 (13)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 14 (21) | 7 (8)
Oral pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 6 (8) | 6 (10)
Vomiting (Gastrointestinal disorders) | 14 (21) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal failure (Renal and urinary disorders) | 3 (3) | 4 (4) — Registered as "Renal failure acute" (in Intuvax [INN: ilixadencel] group, 1 subject [1 unique event], in sunitinib-only group, 2 subjects [2 unique events]) and "Renal failure chronic" (in each group, 2 subjects are affected by 2 unique events)
Renal impairment (Renal and urinary disorders) | 2 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7) | 2 (2)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Hypothyroidism (Endocrine disorders) | 8 (9) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 10 (12) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (6) | 2 (3)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (6) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (8) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 12 (18) | 6 (6)
Hypotension (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of subjects analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT02432846/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT02432846/SAP_001.pdf